CLINICAL TRIAL: NCT02144324
Title: A Comparison of the Skeletal and Dento-alveolar Changes After Treatment of Class III Malocclusion With a Modified Tandem Appliance Versus the Face Mask
Brief Title: Changes Following the Treatment of Lower Jaw Protrusion Using Two Appliances
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Damascus University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UDDS-Ortho-01-2014
Record Dates: First submitted 2014-05-16; First posted 2014-05-22 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Class III Malocclusion in Growing Patients
Keywords: Maxillary protraction; Modified Tandem Appliance; Face mask therapy; Class III malocclusion; Maxillary deficiency
MeSH Terms: conditions — Malocclusion, Angle Class III; Retrognathia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Tandem Appliance (Experimental): This group of patients will receive the new appliance which is called the Tandem Appliance
  Interventions: Device: Tandem Appliance
- Traditional Treatment (No Intervention): Patients in this group will be treated by the traditional Face Mask appliance.

INTERVENTIONS:
Device: Tandem Appliance — We are going to use a modified version of the Tandem Appliance
  Arms: Tandem Appliance

SUMMARY:
An in vivo study evaluating the efficacy of the Tandem appliance in the treatment of maxillary deficiency in growing patients compared to the conventional facemask appliance treatment. Pre-treatment and post-treatment lateral cephalograms will be taken. Dentofacial, sagittal and vertical skeletal measurements will be taken at three assessment times. Changes within each group will be assessed. In addition, the changes between the two groups will be compared.

DETAILED DESCRIPTION:
Maxillary deficiency or retrusion is generally accepted as one of the most difficult and complex orthodontic anomalies to diagnose and treat. Facemask therapy is usually preferred for the treatment of subjects with skeletal and dental Class III malocclusions with a retruded maxilla, and it is known that if the patient is sufficiently motivated to wear a facemask, this type of therapy is quite successful. patient compliance required during facemask therapy due to its poor aesthetics and intraoral appliances for Class III malocclusion treatment such as the Fränkel III , bionator III don't give treatment goals .Hybrid appliance tandem traction bow appliance (TTBA)is introduced by Chun et al. 1999 , as a more aesthetic, effective and comfortable device. Klempner, 2003 modified tandem appliance and published two case reports suggested that TTBA and modified applications have a similar treatment effect to that of an expander-facemask combination(2). A review of the literature showed that there were no statistical studies documenting the effects of modified tandem appliance comparing to traditional expander-facemask therapy and these are the investigators study purposes.

Study design: patients aged between 8-10 with anterior cross bite will be selected from orthodontic department in faculty of dentistry in Damascus university. Pretreatment cephalometric radiography will be taken. Subjects follow inclusion criteria (Skeletal Class III (ANB < 0 degree), due to maxillary retrusion, or a combination of maxillary retrusion and mandibular protrusion, Angle Class III malocclusion with an anterior crossbite., an optimum SN/GoGn angle between 26 and 38 degrees ,fully erupted maxillary incisors,,no congenitally missing teeth or congenital syndromes such as a cleft lip/palate will be . Patient will divided to two group tandem group and face mask group depended on growth pattern. Where from patients in face mask group have normal or horizontal growth pattern,tandem group have vertical one.

Appliance Design The Tandem Appliance comprises three separate components,two fixed and one removable. The upper section is a fixed McNamara expander with buccal arms soldered for attachment of protraction elastics. The lower section is consist of two bands with buccal headgear tubes and buccolingual welded arch for support . Third one is head-gear facebow inserted into the lower tubes and the outer bows bent out for elastics attachment. At the beginning of treatment, patients or Panther are instructed to wear the appliance with light, 8oz /14-16/ hours a day training elastics from the outer face-bow to the buccal arms of the upper expander. Subsequently, heavy orthopedic traction with 14oz /14-16/ hours a day,elastics effectively delivers the protraction force to the maxilla. Lateral cephalometric radiographs without the expander will be taken after a Class I molar relationship and a minimum overjet of 2 mm is obtained. Pre-treatment and post-treatment lateral cephalmetric dentofacial , sagittal and vertical skeletal parameters will be retraced by the author . Statistical analysis will be undertaken using the Statistical Package for Social Sciences, Windows version 19.0 (SPSS Inc., Chicago, Illinois, USA) Paired t-test will be used to evaluate the treatment effects and changes in same group. In depended t-test will be used to evaluate the treatment effects I between groups. confidence level 95% (P< 0.05).

ELIGIBILITY:
Inclusion Criteria:

1. Skeletal Class III (ANB angle < 0 degree) with due to maxillary retrusion, or a combination of maxillary retrusion and mandibular protrusion.
2. Angle Class III malocclusion with an anterior crossbite.
3. An optimum SN/GoGn angle (between 26 and 38 degrees).
4. Fully erupted maxillary incisors.

Exclusion Criteria:

1. Congenitally missing teeth or congenital syndromes such as a cleft lip/palate
2. History of previous orthodontic treatment

Ages: 8 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2014-05; Primary Completion 2015-03 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Change in the SNA angle | This variable will be measured twice: (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment.
  This variable is measured on the lateral cephalogram taken at two time points. This variable is used to give an information about the relative position of the upper jaw in relation to the anterior cranial base.
Change in the spatial position of Point A | This variable will be measured twice: (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment.
  Point A is defined as the point at the maximum concavity of the anterior upper alveolus (containing the upper incisors). The horizontal distance between Point A and the N-perpendicular will be also used to determine the antero-posterior positioning of Point A before and after treatment

SECONDARY OUTCOMES:
Change in the SNB angle | This variable will be measured twice: (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment.
  B is a point located on the mandible on the lateral cephalogram This point is used to determine the antero-posterior positioning of the mandible (lower jaw).
Change in the overjet value | This variable will be measured twice: (T1) baseline measurement at seven days before the beginning of treatment and (T2) at seven days following the end of treatment.
  Overjet is defined as the horizontal overlap between the upper an lower anterior teeth. This variable is going to be measured twice in order to see the changes that occurred in each group antero-posteriorly as a result of the provided orthodontic appliance.

CONTACTS AND LOCATIONS:
Overall Officials: Amro Husson, DDS, Principal Investigator — MSc student, Department of Orthodontics, University of Damascus Dental School; Ahamd Burhan, DDS MSc PhD, Study Chair — Senior Lecturer in Orthodontics, University of Al-Baath Dental School, Hamah, Syria
Locations (1):
- Department of Orthodontics, University of Damascus Dental School, Damascus, Rif-dimashq Governorate, Syria

REFERENCES:
- [Background] Atalay Z, Tortop T. Dentofacial effects of a modified tandem traction bow appliance. Eur J Orthod. 2010 Dec;32(6):655-61. doi: 10.1093/ejo/cjp153. Epub 2010 Mar 26. PMID 20348164
- [Background] Chun YS, Jeong SG, Row J, Yang SJ. A new appliance for orthopedic correction of Class III malocclusion. J Clin Orthod. 1999 Dec;33(12):705-11. No abstract available. PMID 10895664
- [Background] Klempner LS. Early orthopedic Class III treatment with a modified tandem appliance. J Clin Orthod. 2003 Apr;37(4):218-23; quiz 204. No abstract available. PMID 12747076
- [Background] Klempner L. Early treatment of skeletal Class III open bite with the Tandem Appliance. J Clin Orthod. 2011 Jun;45(6):308-16; quiz 339. No abstract available. PMID 21778583
- [Derived] Owens D, Watkinson S, Harrison JE, Turner S, Worthington HV. Orthodontic treatment for prominent lower front teeth (Class III malocclusion) in children. Cochrane Database Syst Rev. 2024 Apr 10;4(4):CD003451. doi: 10.1002/14651858.CD003451.pub3. PMID 38597341